CLINICAL TRIAL: NCT01623713
Title: A Randomized, Double-Blind, Active-Controlled, Multicenter Study to Evaluate Efficacy and Safety Study of Iloperidone Virus Risperidone to Treat Schizophrenia
Brief Title: Efficacy and Safety Study of Iloperidone Virus Risperidone to Treat Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YPLT20111123
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia; Iloperidone; Efficacy
Keywords: schizophrenia; iloperidone; Risperidone; Efficacy; Safety
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone (Active Comparator)
  Interventions: Drug: Risperidone
- iloperidone (Experimental)
  Interventions: Drug: iloperidone

INTERVENTIONS:
Drug: iloperidone — Iloperidone is being development as a treatment of schizophrenia. This trial will verify the safety and efficacy of iloperidone in patients with schizophrenia.
  Arms: iloperidone
Drug: Risperidone — Risperidone is used for the treatment of schizophrenia.Risperidone is unique among most other atypicals in that it has high affinity for the D2 receptor whereas most other atypicals have 'loose binding' of the D2 receptor. It has actions at several 5-HT (serotonin) receptor subtypes.
  Arms: Risperidone

SUMMARY:
The purpose of this study is to determine whether iloperidone is effective in the treatment of Schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 18-65 years old.
* DSM-IV diagnosis of schizophrenia.
* PANSS≥70.
* Of the 7 PANSS positive symptom subscale, at least two score ≥ 4 points.
* Written informed consent.

Exclusion Criteria:

* Pregnant or nursing (lactating) women, or women who plan on conceiving during the course of the study.
* Clinically significant disease of the heart,kidneys,liver,hematonosis or endocrine system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale(PANSS)-Total Score | 6 weeks

SECONDARY OUTCOMES:
Effective percentage(PANSS score reduce rate≥50%) | 6 weeks
Change in scores from baseline to end point assessment on the PANSS Positive subscale (PANSS-P) | 6 weeks
Change in scores from baseline to end point assessment on the PANSS Negative subscale (PANSS-N) | 6 weeks
Change in scores from baseline to end point assessment on the PANSS General Psychopathology subscale(PANSS-GP) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Hospital of Peking University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203